CLINICAL TRIAL: NCT01215708
Title: Effect of Tamsulosin and Nifedipine on the Elimination of Fragments After Extracorporeal Shock Waves Lithotripsy in Patients With Kidney Stones - a Prospective, Double-blind and Randomized Study
Brief Title: Effects of the Use of Adjuvant Drugs After Extracorporeal Shockwave Lithotripsy (ESWL) in Renal Calculus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Fabio Carvalho Vicentini, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 278/06
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-09

CONDITIONS: Renal Calculi
Keywords: Kidney calculi; Lithotripsy; Calcium channel blockers; Adrenergic alpha-antagonists.
MeSH Terms: conditions — Kidney Calculi | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nifedipine (Active Comparator): nifedipine retard 20mg daily
  Interventions: Drug: Tamsulosin
- tamsulosin (Active Comparator): tamsulosin 0,4mg
  Interventions: Drug: Tamsulosin
- placebo (Placebo Comparator): placebo capsule
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — tamsulosin 0,4mg every night for 30 consecutive days
  Other Names: secotex

SUMMARY:
The investigators objective is to study if some drugs can improve the success rate of extracorporeal shockwave lithotripsy for renal stones.

DETAILED DESCRIPTION:
Extracorporeal shockwave lithotripsy is one of the modalities of treatment of renal stones. It´s a machine that breaks the renal stones extracorporeally. Some drugs, like alpha blockers and calcium channel blockers, can improve the success rates of this procedure. Our objective is to study the real effects of two drugs, tamsulosin and nifedipine, compared to placebo, in the elimination of fragments after the extracorporeal shockwave lithotripsy treatment.

ELIGIBILITY:
Inclusion Criteria:

* radiopaque renal stone, 5 to 20 mm, located at renal pelvis or superior or middle calix

Exclusion Criteria:

* inferior calix, any contraindication for extracorporeal shockwave lithotripsy, pregnancy, coagulopathy, previous renal surgery, age under 18, abdominal aorta aneurism and urinary infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-08; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of Tamsulosin and Nifedipine in the success rates after treatment of radiopaque renal stones between 5-20 mm with only one session of SWL | 30 days

SECONDARY OUTCOMES:
To evaluate the effects of Tamsulosin and Nifedipine in the episodes of pain after treatment of radiopaque renal stones between 5-20 mm with only one session of SWL | 30 days
To evaluate the effects of Tamsulosin and Nifedipine in the velocity of elimination of fragments after treatment of radiopaque renal stones between 5-20 mm with only one session of SWL | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Srougi, MD, Study Chair — University of Sao Paulo
Locations (1):
- Clinics Hospital of University of Sao Paulo, São Paulo, São Paulo, Brazil